CLINICAL TRIAL: NCT01018069
Title: An Open-Label Randomized Phase 2 Study of the X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 Given in Combination With High-dose Cytarabine and Idarubicin in AML Following Failure of a Single Standard Dose Cytarabine Based Frontline Induction Regimen
Brief Title: AEG35156 in Combination With High-dose Cytarabine and Idarubicin in AML Following Failure of a Single Standard Dose Cytarabine Based Frontline Induction Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failed to reach endpoints
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, Aegera Therapeutics Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-206; 2009-013669-25 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Leukemia
Keywords: Acute; myeloid; leukemia; antisense; chemotherapy; idarubicin; cytarabine; Patients with AML, except those with APL (acute promyelocytic leukemia), failing a single standard dose cytarabine based frontline induction regimen.
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — AEG 35156

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AEG35156 (Active Comparator): Patient receive AEG35156 prior to chemotherapy
  Interventions: Drug: AEG35156
- Control (Sham Comparator): Patients receive chemotherapy only
  Interventions: Drug: AEG35156

INTERVENTIONS:
Drug: AEG35156 — 2 hr infusion of 650 mg of AEG35156 on days 1, 2, 3 and 8. Idarubicin 12 mg/m2 over 30 minutes daily on each of days 4, 5 and 6. The dose of cytarabine will be 1.5 g/m2 daily by continuous infusion x 4 days (days 4-7) in patients under age 65 and x 3 days (days 4-6) in patients age 65 and above.

SUMMARY:
To determine if AEG35156 can enhance the combined complete remission (CR) and CR with incomplete platelet recovery (CRp) rate of high-dose cytarabine and idarubicin in AML following failure of a single standard dose cytarabine based frontline induction regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, except those with APL (acute promyelocytic leukemia), failing a single standard dose cytarabine based frontline induction regimen. The diagnosis of refractory AML is based on the presence of either > 10% blasts in marrow or blood or 5-10% blasts in either site together with cytopenia (Hb < 10 g/dL, or platelets < 100 x 109/L, or neutrophil count < 1.0 x 109/L).
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Male, or female patients who are post-menopausal (amenorrheic for at least 12 months), or surgically or biologically sterile.
* Patients must have adequate organ and immune function as indicated by the following laboratory values:

Parameter Laboratory Values Serum creatinine; ≤2.0 mg/dL (≤ 177 μmol/L Total Bilirubin ≤2.0 mg/dL (≤ 34 μmol/L) AST (SGOT) and ALT (SGPT) ≤3 X ULN

* The patient must understand, be able and willing and likely to fully comply with study procedures, including scheduled follow-up, and restrictions.

Exclusion Criteria:

* Clinical evidence of ongoing grade 3 or 4 non-hematological toxicities from the initial standard dose cytarabine-based induction chemotherapy
* Patients with a prior history of peripheral neuropathy of grade 2 or higher.
* Clinical evidence of active CNS leukemic involvement.
* Active and uncontrolled infection. Patients with an infection who are under active treatment with antibiotics and whose infections are controlled may be entered to the study.
* Current evidence of invasive fungal infection (blood or tissue culture).
* Current evidence of an active second malignancy except for non-melanoma skin cancer.
* Uncontrolled medical problems, unrelated to the malignancy, or of sufficient severity that in the opinion of the investigator, impair a patient's ability to give informed consent or unacceptably reduce the safety of the proposed treatment.
* Neurological or psychiatric disorders that would interfere with consent or study follow-up.
* Known or suspected intolerance or hypersensitivity to the study drugs [or closely related compounds] or any of their stated ingredients. Study drugs being the antisense, cytarabine and idarubicin.
* History of alcohol or other substance abuse within the last year.
* Use of another investigational agent within the last 14 days prior to enrolment. Patients who have received a previous antisense agent in the last 90 days will be excluded.
* Female patients who are pregnant, lactating, or with a positive pregnancy test at screening must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine if AEG35156 can enhance the CR and CR with incomplete platelet recovery (CRp) rate and duration of high-dose cytarabine and idarubicin in AML following failure of a single standard dose cytarabine based frontline induction regimen. | 1 year

SECONDARY OUTCOMES:
To determine if AEG35156 can enhance overall survival, is safe and measured (Pharmacokinetic) following high-dose cytarabine and idarubicin in AML following failure of a single standard dose cytarabine based frontline induction regimen. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Schimmer, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (18):
- United States (6):
  - UCLA School of Medicine, Los Angeles, California
  - Rocky Mountain Blood & Marrow Transplant Program, Denver, Colorado
  - Northwestern University Med School, div. Oncology & Hematology, Chicago, Illinois
  - New York Medical College, Valhalla, New York
  - MD Anderson Cancer Center University of Texas, Houston, Texas
  - Cancer Research Institute of Scott & White Hospital, Temple, Texas
- Canada (4):
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
- Germany (8):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - St. Johannes Hospital, Duisburg
  - Universitatsklinimum Essen, Essen
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - 2. Medizinische Klinik und Poliklinik im Stadtischen Krankenhaus Kile GmgH, Kiel
  - III. Medizinische Klinik und Poliklinik der Johannes Gutenberg-Universitat, Mainz
  - Medizinische Klinik a Hamatologie und Onkologie, Münster
  - Robert Boasch Krankenhaus Stuttgart, Stuttgart